CLINICAL TRIAL: NCT05234788
Title: Renal Artery DenervatIon Using Radial accesS in Uncontrolled HyperTensioN:Non Inferiority Study Comparing Safety and Efficacy of Radio Frequency Renal Denervation Using Iberis Renal Denervation System Via Radial Access Compared With Femoral
Brief Title: Renal Artery DenervatIon Using Radial accesS in Uncontrolled HyperTensioN
Acronym: RADIUS-HTN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai AngioCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-01
Record Dates: First submitted 2022-01-06; First posted 2022-02-10 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
Keywords: Renal Denervation; TransRadial; Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TransRadial access (Experimental): Patients in this group are thus treated using a TRA approach
  Interventions: Procedure: Transradial Renal Denervation
- TransFemoral Access (Active Comparator): Patients in this group are thus treated using a TFA approach.
  Interventions: Procedure: Transfemoral Renal Denervation

INTERVENTIONS:
Procedure: Transfemoral Renal Denervation — Radiofrequency renal denervation using the Iberis Renal Denervation System treated via femoral artery access
  Other Names: TFA RDN
  Arms: TransFemoral Access
Procedure: Transradial Renal Denervation — Radiofrequency renal denervation using the Iberis Renal Denervation System treated via radial artery access
  Other Names: TRA RDN
  Arms: TransRadial access

SUMMARY:
Non-inferiority, prospective, multi-center, international, post-market, randomized (1:1) clinical trial in patients with uncontrolled hypertension to compare the safety and efficacy of radio frequency renal denervation using Iberis Renal Denervation System via radial access compared with femoral access.

DETAILED DESCRIPTION:
Non-inferiority, prospective, multi-center, international, post-market, randomized (1:1) clinical trial.

90 patients with uncontrolled hypertension treated with 2 to 5 antihypertensive drugs including one angiotensin receptor blocker (ARB) or angiotensin-converting enzyme Inhibitor (ACE-I) in combination with one diuretic or calcium channel blocker will be randomized in a 1:1 ratio to the radial access renal denervation group (intervention) or the femoral access renal denervation group (control).

Around 12 sites in 3 European countries (France, Germany and Switzerland) are planned to enroll 90 patients.

For patients with a contraindication for the TransFemoral Access (major femoral disease, bilateral femoral vascular prosthesis, extreme obesity), a register is also carried out in parallel with the study. The inclusion and exclusion criteria will be the same except the fact that patients have to be eligible for TransFemoral access, endpoints and data collected will be the same.

All patients will be followed per standard of care practice and follow-up visits are scheduled at 3 months (follow-up time window +14 days) and 6 months (follow-up time window +30 days).

Estimated duration of inclusions: 27 months. Total estimated duration of study: 38 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 and ≤75 years old
2. Persistent uncontrolled hypertension defined as the mean of three consecutive measurements of systolic office blood pressure >150 mmHg and diastolic office blood pressure >80 mmHg as well as ambulatory daytime systolic blood pressure ≥140 mmHg despite prescription of 2 to 5 anti-hypertensive drugs including an angiotensin-receptor blocker or an angiotensin-converting enzyme inhibitor in combination with a diuretic or calcium channel blocker
3. Renal artery diameter ≥3 mm and ≤8 mm (to be assessed during the procedure)
4. Patient can be treated according to the instructions for use (IFU)
5. Patient eligible for TransFemoral Access and TransRadial Access
6. Patient, who understands the trial requirements and the treatment procedures and provides written informed consent

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) <45 mL/min/m² (MDRD formula)
2. Prior renal transplant
3. Presence of accessory artery (polar artery) supplying more than 20% of renal parenchyma that cannot be treated (renal artery diameter <3 mm) with renal denervation
4. Patient lacking capacity (i.e. patient suffering from dementia and others) to provide informed consent
5. Patient currently participating in another investigational drug or device study
6. Pregnant or breastfeeding women or those intending to become pregnant before the end of the follow-up
7. Subjects under judicial protection, guardianship or curatorship or subjects deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in office systolic blood pressure at 3 months. | 3 months
  Mean of 3 readings at 1-minute intervals after a 5-minute resting period in the examination room (mmHg)

SECONDARY OUTCOMES:
Procedural success | Procedure
  Number of participants with successful completion of the renal denervation procedure via the intended approach
Number of ablations per patient | Procedure
  Number of ablations performed during the procedure for each participants
Procedural duration | Procedure
  Lenght of the procedure
X-Ray exposure | Procedure
  Level of X-Ray exposure
Volume of contrast media | Procedure
  Volume of contrast media use during the procedure
Major vascular events | Discharge or at least 24hours after procedure)
  major hematoma, pseudoaneurysm, arteriovenous fistula, retroperitoneal hematoma, arterial thrombosis, dissection and perforation, distal embolization, femoral nerve injury, local infection and arterial avulsion
Office systolic blood pressure | 6 months
  Mean of 3 readings at 1-minute intervals after a 5-minute resting period in the examination room (mmHg)
Office diastolic blood pressure | 3 months and 6 months
  Mean of 3 readings at 1-minute intervals after a 5-minute resting period in the examination room (mmHg)
Mean 24-hour ambulatory systolic and diastolic blood pressure | 3 months and 6 months
Daytime (7:00 am to 10:00 pm) and nighttime (10:00 pm to 7:00 am) ambulatory systolic and diastolic blood pressure | 3 months and 6 months
  Mean (mmHg)
Percentage of patients at target blood pressure | 3 months and 6 months
Office heart rate | 3 months and 6 months
  beats per minute
Ambulatory heart rate | 3 months and 6 months
  beat per minute
Home blood pressure | 7 days prior to baseline/randomization and before every follow-up
  3 measurements in the morning and evening for 7 days
Home heart rate | 7 days prior to baseline/randomization and before every follow-up
  3 measurements in the morning and evening
Renal function | 3 months and 6 months
  change of estimated-Glomerular Filtration Rate (eGFR)
Renal artery safety | 6 months
  absence of renal re-intervention, renal artery stenosis or dissection.
Changes in medication (DDD Defined Daily Doses) | 3 and 6 months
Length of in-hospital stay | Discharge (up to 48 hours)
Percentage of Vascular Access Site Complication (VASC) | Discharge (up to 48 hours), 3 and 6 months
Percentage of stroke / TIA | Discharge (up to 48 hours), 3 and 6 months
  Percentage of stroke and/or transient ischemic attack
Percentage of Bleeding | Discharge (up to 48 hours), 3 and 6 months
  Percentage of bleeding (BARC 3 to 5)
Patient satisfaction | Discharge (up to 48 hours) and 3 months
  Assessed by the Medical Outcomes Study Short Form 36-item health status questionnaire (acute SF-36) and a series of procedure-specific questions
Time in target range | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, MD, MA, Principal Investigator — University Hospital, Basel, Switzerland
Locations (11):
- France (4):
  - Hôpital Saint André, Bordeaux
  - Hôpital Jacques Cartier, Massy
  - Centre Hospitalier de Pau, Pau
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden Neustadt GbR, Dresden
  - Asklepios Klinik Altona, Hamburg
  - Saarland University Hospital, Homburg
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal
- Switzerland (3):
  - University Hospital Basel, Basel
  - University & Hospital Fribourg, Fribourg
  - Cardiovascolare Istituto Cardiocentro Ticino, Lugano